CLINICAL TRIAL: NCT00985062
Title: Food Lifestyle and Fertility Outcome
Brief Title: Mild Versus Conventional Ovarian Stimulation Treatment for In Vitro Fertilization
Acronym: FOLFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Dr. R.P.M. Steegers-Theunissen, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VPG.03.02
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Subfertility
Keywords: Folic Acid; Homocysteine; Ovarian response; In Vitro Fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mild Ovarian Stimulation (Active Comparator)
  Interventions: Procedure: Mild Ovarian Stimulation Treatment
- Conventional Ovarian Stimulation (Active Comparator)
  Interventions: Procedure: Conventional Ovarian Stimulation Treatment

INTERVENTIONS:
Procedure: Mild Ovarian Stimulation Treatment — Administration of a fixed dose of 150 IU/day rFSH s.c. (Puregon® NV Organon, Oss, The Netherlands) from cycle day 5 onwards. As soon as the leading follicle reached a diameter of 14mm, a GnRH-antagonist (Orgalutran®, NV Organon, Oss, The Netherlands) was administered at 0.25 mg/day s.c.. To induce final oocyte maturation a single s.c. dose of 10.000 IE hCG (Pregnyl®, NV Organon. Oss, The Netherlands) was administered.
  Arms: Mild Ovarian Stimulation
Procedure: Conventional Ovarian Stimulation Treatment — Administration of GnRH agonist Triptorelin (Decapeptyl®, Ferring BV, Hoofddorp, The Netherlands) at 0.1 mg/day s.c., starting on cycle day 21 of the menstrual cycle preceding the actual stimulation cycle. After two weeks of the GnRH regimen, co-treatment with rFSH 225 IU/day s.c. (Puregon®, NV Organon, Oss, The Netherlands) was initiated. To induce final oocyte maturation a single s.c. dose of 10.000 IE hCG (Pregnyl®, NV Organon. Oss, The Netherlands) was administered
  Arms: Conventional Ovarian Stimulation

SUMMARY:
In vitro fertilization (IVF) is an assisted reproductive technique to achieve pregnancy in subfertile couples of which the average success rate is only 25%. Mild ovarian stimulation treatment yields less oocytes, has less adverse effects but has a comparable clinical outcome compared to conventional stimulation treatment. There is high inter- and intra person variability in ovarian response and fertility outcome parameters after stimulation treatment and little is known about explanatory variables herefore.

Nutrition and in particular folate, or its synthetic derivative folic acid, is a B-vitamin which has been widely asssociated with reproductive outcome and subfertility. Therefore, in this study we aim to investigate the influence of preconception nutrition and folic acid use on ovarian response after mild/conventional stimulation treatment and to identify biomarkers in the follicular fluid which can indicate oocyte quality and other fertility outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All couples with an indication for IVF/ICSI treatment in the Erasmus Medical Center

Exclusion Criteria:

* Prior oocyte donation
* Endometriosis
* Hydrosalpinx
* MESA/PESA
* Age >37
* BMI <18 or >29kg/m2
* Menstrual cycle disruptions
* Indication for Intra Cytoplasmic Sperm Injection (ICSI)
* Prior IVF treatment without embryo transplant
* History of recurrent abortion
* Abnormal karyotype of male/female
* Uterine abnormalities

Max Age: 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2004-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Endocrine, metabolic biomarkers and proteins and Fertility outcome parameters | At menstrual cycle day 2 before stimulation, on the day of hCG administration after stimulation treatment and after embryo transplantation

SECONDARY OUTCOMES:
Homocysteine-methionine cycle biomarker, endocrine and folate levels in serum | At menstrual cycle day 2 before stimulation and on the day of hCG administration after stimulation treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Forges T, Pellanda H, Diligent C, Monnier P, Gueant JL. [Do folates have an impact on fertility?]. Gynecol Obstet Fertil. 2008 Sep;36(9):930-9. doi: 10.1016/j.gyobfe.2008.07.004. Epub 2008 Aug 12. French. PMID 18701335
- [Background] Fauser BC, Diedrich K, Devroey P; Evian Annual Reproduction Workshop Group 2007. Predictors of ovarian response: progress towards individualized treatment in ovulation induction and ovarian stimulation. Hum Reprod Update. 2008 Jan-Feb;14(1):1-14. doi: 10.1093/humupd/dmm034. Epub 2007 Nov 15. PMID 18006561
- [Background] Verberg MF, Eijkemans MJ, Macklon NS, Heijnen EM, Baart EB, Hohmann FP, Fauser BC, Broekmans FJ. The clinical significance of the retrieval of a low number of oocytes following mild ovarian stimulation for IVF: a meta-analysis. Hum Reprod Update. 2009 Jan-Feb;15(1):5-12. doi: 10.1093/humupd/dmn053. PMID 19091754
- [Background] Verberg MF, Macklon NS, Nargund G, Frydman R, Devroey P, Broekmans FJ, Fauser BC. Mild ovarian stimulation for IVF. Hum Reprod Update. 2009 Jan-Feb;15(1):13-29. doi: 10.1093/humupd/dmn056. PMID 19091755
- [Result] Baart EB, Martini E, Eijkemans MJ, Van Opstal D, Beckers NG, Verhoeff A, Macklon NS, Fauser BC. Milder ovarian stimulation for in-vitro fertilization reduces aneuploidy in the human preimplantation embryo: a randomized controlled trial. Hum Reprod. 2007 Apr;22(4):980-8. doi: 10.1093/humrep/del484. Epub 2007 Jan 4. PMID 17204525